CLINICAL TRIAL: NCT05756439
Title: Hemodynamic Changes During Implant Surgery with Intravenous Conscious Sedation: a Clinical Prospective Study
Brief Title: Hemodynamic Changes During Implant Surgery with Intravenous Conscious Sedation
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hom-Lay Wang, DDS, MSD, Ph D, Collegiate Professor of Periodontics and Professor of Dentistry, University of Michigan
Other Study IDs: HUM00172521
Record Dates: First submitted 2023-02-02; First posted 2023-03-06 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2023-02

CONDITIONS: Blood Pressure; Dental Anxiety
Keywords: Dental surgery; intravenous sedation
MeSH Terms: interventions — Analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: Participants having dental surgery
  Interventions: Drug: No IV sedation
- Intravenous sedation: Participants having dental surgery
  Interventions: Drug: Intravenous Sedatives with or Without Analgesia

INTERVENTIONS:
Drug: Intravenous Sedatives with or Without Analgesia — Participants having dental surgery with conscious intravenous sedation
  Other Names: conscious iv sedation
  Groups: Intravenous sedation
Drug: No IV sedation — Participants having dental surgery without conscious intravenous sedation
  Other Names: no conscious iv sedation
  Groups: Control

SUMMARY:
The goal of this study is to determine whether intravenous sedation would contribute to the stabilization of hemodynamics in adult patients during periodontal/implant surgery compared to receiving local anesthesia during periodontal/implant surgery

DETAILED DESCRIPTION:
Monitoring is the global method of observation and data recording in relation to body organ and system function that afford constant information to ensure continuous evaluation of the patient's physical condition. The aim of this study is to determine whether intravenous sedation would contribute to the stabilization of hemodynamics in adult patients during dental surgery.

Secondary, patient related outcome will be evaluated by a questionnaire to determine the patients' perception, acceptance and comfort during intravenous sedation after assessing the influence of patients' preoperative anxiety.

50 subjects who need implant/periodontal surgery at the University of Michigan School of Dentistry will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 18 years of age
* Need dental implant/periodontal surgery with or without IV sedation (up to a maximum of 4 implants)

Exclusion Criteria:

* You have any reason you cannot comply with the study protocol
* You take any medication that may influence hemodynamic changes including anxiolytic medication (last intake <48 hours before intervention) as well as pain medication (last intake <48 hours before intervention)
* Pregnant or unsure of pregnancy (self-reported)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects scheduled for dental surgery with or without intravenous sedation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure (systolic) | At the start of surgery and every 15 minutes until the surgery is over, up to 4 hours.
  Systolic blood pressure will be recorded throughout the surgical procedure
Change in blood pressure (diastolic) | At the start of surgery and every 15 minutes until the surgery is over, up to 4 hours.
  Diastolic blood pressure will be recorded throughout the surgical procedure
Change in heart rate | At the start of surgery and every 15 minutes until the surgery is over, up to 4 hours.
  Heart rate will be recorded throughout the surgical procedure
Change in oxygen saturation | At the start of surgery and every 15 minutes until the surgery is over, up to 4 hours.
  Oxygen saturation will be recorded throughout the surgical procedure

SECONDARY OUTCOMES:
Dental Anxiety Scale | Baseline
  Evaluation of dental anxiety using Corah's Dental Anxiety Scale. Minimum score 4, maximum score 20 with higher scores indicating greater dental anxiety.
Patient Satisfaction | 2 weeks after surgery
  Patient satisfaction with surgery. Minimum score 6, maximum score 30 with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Hom-Lay Wang, DDS MSD PhD, Principal Investigator — Department of Periodontics and Oral Medicine University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States